CLINICAL TRIAL: NCT06618287
Title: A Phase 1/2a, Open-label, Dose-finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BMS-986507 (BL-B01D1) Combinations in Adult Participants With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Preliminary Efficacy of BMS-986507 Combinations in Adult Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA244-0001; 2024-514947-27 (Other: EU CTR); U1111-1308-2752 (Other: WHO)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Breast Cancer
Keywords: Non-Small Cell Lung Cancer (NSCLC); Epidermal Growth Factor Receptor mutated (EGFRmt); Epidermal Growth Factor Receptor wild-type (EGFRwt); Triple-negative breast cancer (TNBC)
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — osimertinib; pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental)
  Interventions: Drug: BMS-986507; Drug: Osimertinib
- Group B (Experimental)
  Interventions: Drug: BMS-986507; Drug: Pembrolizumab
- Group C (Experimental)
  Interventions: Drug: BMS-986507; Drug: Nivolumab
- Group D (Experimental)
  Interventions: Drug: BMS-986507; Drug: Pumitamig
- Group E (Experimental)
  Interventions: Drug: BMS-986507; Drug: Pumitamig

INTERVENTIONS:
Drug: BMS-986507 — Specified dose on specified days
  Other Names: Iza-bren; Izalontamab brengitecan
Drug: Osimertinib — Specified dose on specified days
  Arms: Group A
Drug: Pembrolizumab — Specified dose on specified days
  Arms: Group B
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Group C
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545; BNT327; PM8002
  Arms: Group D; Group E

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, and preliminary efficacy of BMS-986507 combinations in adult participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Participants must have at least one measurable lesion per response evaluation criteria in solid tumors.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Participants must have a life expectancy of at least 3 months at the time of the first dose.
* Group A: Participants must have pathologically confirmed locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation in exon 21, either alone or in combination with other EGFR mutations, which may include T790M in exon 20. Participants with other EGFR mutations (including but not limited to, exon 21 L861Q, exon 18 G719X, and exon 20 S768I mutations, etc.) will also be allowed
* Group B: Participants must have pathologically confirmed locally advanced or metastatic NSCLC.
* Group C: Participants must have pathologically confirmed locally-advanced, recurrent inoperable, or metastatic TNBC or ER-low, HER2-negative BC.
* Group D: Participants must have pathologically confirmed locally-advanced, recurrent inoperable, or metastatic TNBC per ASCO/CAP criteria, based on the most recently analyzed biopsy or another pathology specimen.
* Group E: Participants must have pathologically confirmed locally advanced or metastatic NSCLC, not amenable to treatment in curative intent.

Exclusion Criteria

* Participants must not have any mixed Small Cell Lung Cancer (SCLC) and Non-Small Cell Lung Cancer (NSCLC) histology.
* Participants with known mutations in EGFR will be excluded (Group A,B and E).
* Participants must not have a history of serious recurrent infections.
* Participants must not have a history of severe heart disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2031-02-26 (Estimated); Study Completion 2031-02-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 3 years
Number of participants with serious adverse events (SAEs) | Up to 3 years
Number of participants with AEs meeting protocol defined dose-limiting toxicity (DLT) critera | Up to 3 years
Number of participants with AEs leading to discontinuation | Up to 3 years
Number of participants with AEs leading to death | Up to 3 years
Number of DLTs that occur during the DLT evaluation period | Up to 3 weeks

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 3 years
Time of maximum observed concentration (Tmax) | Up to 3 years
Area under the concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to 3 years
Area under the serum concentration-time curve within a dosing interval (AUC(TAU)) | Up to 3 years
Objective response rate (ORR) | Up to 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (56):
- United States (12):
  - Local Institution - 0066, Birmingham, Alabama
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Local Institution - 0065, Iowa City, Iowa
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 0102, Columbus, Ohio
  - Local Institution - 0052, Portland, Oregon
  - Local Institution - 0090, Portland, Oregon
  - Local Institution - 0014, Pittsburgh, Pennsylvania
  - Local Institution - 0103, Knoxville, Tennessee
  - Local Institution - 0092, Irving, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Local Institution - 0064, Newmarket, Ontario
  - Local Institution - 0023, Ottawa, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Chile (5):
  - Local Institution - 0105, Valdivia, Los Ríos Region
  - Local Institution - 0107, Viña del Mar, Región de Valparaíso
  - Local Institution - 0048, Santiago, Santiago Metropolitan
  - Local Institution - 0049, Santiago, Santiago Metropolitan
  - Local Institution - 0047, Santiago, Santiago Metropolitan
- France (9):
  - Local Institution - 0077, Nice, Alpes-Maritimes
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier, Hérault
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Local Institution - 0076, Caen
  - Institut Curie, Paris
  - Hôpital Tenon, Paris
- Italy (6):
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Local Institution - 0033, Milan, Lombardy
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Local Institution - 0035, Florence, Tuscany
  - Local Institution - 0093, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Nederlands Kanker Instituut Antoni van Leeuwenhoek (NKI AVL), Amsterdam
- Spain (10):
  - Local Institution - 0062, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, Hospitalet, Barcelona [Barcelona]
  - Local Institution - 0059, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Local Institution - 0061, Majadahonda, Madrid, Comunidad de
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - Royal Free Hospital, London, England
  - Local Institution - 0021, Glasgow, Glasgow City
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Local Institution - 0001, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06618287.html